CLINICAL TRIAL: NCT04552288
Title: Phase II Study of IL-5-receptor-alpha-chain (IL-5Rα) Inhibition With Benralizumab for Eosinophil-Related Cutaneous Adverse Events in Cancer Patients
Brief Title: Study of Benralizumab in People With Skin Side Effects Caused by Cancer Therapies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-344
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Solid Carcinoma; Solid Tumor, Adult; Hematologic Malignancy
Keywords: Benralizumab; hematologic cancer; solid cancer; 20-344; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Hematologic Neoplasms | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with eosinophil-related cutaneous events (Experimental): Study participants will have grade 2/3 eosinophil-related cutaneous adverse events
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — All eligible patients will receive a benralizumab dose of 30 mg SC administered by a healthcare provider once every 4 weeks for the first 3 doses, followed by once every 8 weeks for 3 additional doses.

SUMMARY:
The purpose of this study is to find out whether the study drug benralizumab is a safe treatment that can reduce the skin side effects caused by cancer treatment by reducing the level of eosinophils in your blood. Reducing the skin side effects of your cancer treatment may improve quality of life and allow participants to continue to receive their usual cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically confirmed solid or hematologic cancers.

OR

* Patient is receiving alpelisib for PIK3CA-Related Overgrowth Spectrum disorder.
* Female and male aged 18 to 85 years, inclusively, at the time of Week 0/Day 1 of treatment.
* Patients must have a therapy-related CTCAE grade 2/3 (See Appendix A)cutaneous adverse event defined as any cutaneous reaction listed below and blood eosinophil counts of at least .3 K/mcl.

  * Rash maculo-papular
  * Bullous dermatitis
  * Pruritus
  * Urticaria
  * Eczema
* Patients must plan to continue on culprit drugs (cancer patients).
* Patients planning to receive alpelisib indicated for PIK3CA-Related Overgrowth

Spectrum disorder OR patients receiving immunotherapy and/or targeted therapy, including but not limited to the following agents, will be eligible for inclusion:

* Immunotherapies: ipilimumab, nivolumab, pembrolizumab, avelumab, durvalumab, atezolizumab tremelimumab.
* Targeted therapies: trastuzumab, pertuzumab, alpelisib, osimertinib, everolimus, temsirolimus, sorafenib, regorafenib.

  * Patients using topicals/orals for indication of skin rash/pruritus for at least 7 days should continue using these drugs for the study duration
  * Adequate bone marrow, liver and renal function:
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
* Serum creatinine ≤ 1.8 xULN or calculated creatinine clearance >45 ml/min
* Platelet count > 50 K/mcL , hemoglobin (Hb) > 8 g/dL, absolute neutrophil count (ANC) >1.0 K/mcL. Blood transfusion to meet the inclusion criteria will not be allowed.

  * ECOG performance status 0-1 (see Appendix C).
  * Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
  * Female patients are authorized to participate if they meet the following criteria:
* Women of child bearing potential must meet both of the following conditions:
* Have a negative serum pregnancy test prior to enrollment and within 14 days prior to administration of the investigational product (IP).
* Patient must use an effective form of birth control (confirmed by the Investigator) throughout the study duration and within 16 weeks after last dose of IP.
* Female subjects who cannot bear children as evidenced by one or more of the following:
* Bilateral Oophorectomy
* Bilateral Salpingectomy
* Bilateral Salpingectomy-Oophorectomy
* Hysterectomy
* Menopause (no menses ≥ 1 year prior to treatment)
* Surgical Sterilization (i.e., tubal ligation or blockage) Note: If criteria not met, patient should be regarded as having child bearing potential

  * Subject must be able to receive a subcutaneous injection.
  * New/worsening ercAE within 90 days prior to study enrollment. Note: This assessment will be performed by the treating investigator.

Exclusion Criteria:

* Concurrent use of another investigational drug or device for the ercAE (i.e., outside of study treatment) during, or within 4 weeks of treatment.
* Patients receiving prednisone ≥ 20mg a day.
* Known use of anti-IL-5 agents or biologics for the treatment of asthma which are known to decrease blood eosinophil levels.
* Patients cannot use new topicals or medications for indication of pruritus or skin rash
* Known history of anaphylaxis to biologic therapy.
* A helminthic parasitic infection diagnosed within 24 weeks prior to the first treatment, that had not been treated with, or has failed to respond to, standard of care therapy.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Active infection that would impair the ability of the patient to receive study treatment.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Receipt of live attenuated vaccines 30 days prior to the date of randomization

  ° Receipt of inactive/killed vaccinations (e.g., inactive influenza) is allowed provided they were not administered within 1 week before/after any investigational product administration.
* Known history of allergy or reaction to the investigational product formulation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2026-03-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center Suffolk - Hauppauge (Limited Protocol Activities), Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Eosinophil-related Cutaneous Events
Started | 51
Completed | 14
Not Completed | 37
Not completed — Death | 3
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 9
Not completed — Withdrawal by Subject | 6
Not completed — Disease progression, Complicated disease, Ineligible | 10

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Eosinophil-related Cutaneous Events
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 63 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 38
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in CTCAE Grade 2/3 Eosinophil-related Cutaneous Adverse Events
Description: To evaluate the percent reduction in CTCAE grade 2/3 eosinophil-related cutaneous adverse events to grade ≤1 resulting from checkpoint inhibitors (CPIs) or targeted therapies with absolute blood eosinophil counts of at least .3 K/mcl.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Eosinophil-related Cutaneous Events
Number analyzed (Participants) | 51
Participants
  Participants who responded to treatment | 32
  Participants who did not respond to treatment | 10
  Participants not evaluable | 9

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Participants With Eosinophil-related Cutaneous Events
All-Cause Mortality (participants affected / at risk) | 29/51
Serious Adverse Events (participants affected / at risk) | 4/51
Other Adverse Events (participants affected / at risk) | 37/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Eosinophil-related Cutaneous Events (N=51)
Death - Not other specified (General disorders) | 2
Gastric Perforation (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Eosinophil-related Cutaneous Events (N=51)
Somnolence (Nervous system disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 1
Swelling of gums/lips (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Heart failure (Cardiac disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Pain (General disorders) | 1
Fatigue (General disorders) | 2
Vomiting/Nausea (Gastrointestinal disorders) | 3
Allergic reaction (Immune system disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
EV Rash (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Stomatits (Gastrointestinal disorders) | 3
Elevated liver enzymes (Investigations) | 1
Hypotension (Vascular disorders) | 1
Xerosis (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Edema Limbs (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04552288/Prot_SAP_000.pdf